CLINICAL TRIAL: NCT02938572
Title: Proof-of-Principle Trial Investigating Pharmacodynamics, Pharmacokinetics, and Safety of NNC0143-0406 in Subjects With Type 1 Diabetes Mellitus
Brief Title: A Randomised Proof-of-Principle Trial Investigating Pharmacodynamics, Pharmacokinetics, and Safety of NNC0143-0406 in Subjects With Type 1 Diabetes Mellitus
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: NN1406-4218; 2014-005340-18 (EudraCT Number); U1111-1164-6715 (Other: WHO)
Record Dates: First submitted 2016-10-17; First posted 2016-10-19 (Estimated); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Diabetes; Diabetes Mellitus, Type 1
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1 | interventions — Insulin Aspart

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- NNC0143-0406 (Experimental)
  Interventions: Drug: NNC0143-0406
- Insulin aspart (Active Comparator)
  Interventions: Drug: Insulin Aspart

INTERVENTIONS:
Drug: NNC0143-0406 — Administered subcutaneously (s.c. under the skin)
  Arms: NNC0143-0406
Drug: Insulin Aspart — Administered subcutaneously (s.c. under the skin)
  Arms: Insulin aspart

SUMMARY:
This trial is conducted in Europe. The aim of this trial is to investigate Pharmacodynamics (the effect of the investigated drug on the body) , Pharmacokinetics (the exposure of the trial drug in the body), and Safety of NNC0143-0406 in Subjects with Type 1 Diabetes Mellitus

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-55 years (both inclusive) at the time of signing informed consent
* Subjects diagnosed (clinically) with type 1 diabetes mellitus at least 365 days prior to the day of screening
* Treated with continuous subcutaneous insulin infusion at least 90 days prior to the day of screening

Exclusion Criteria:

* Known or suspected hypersensitivity to trial product(s) or related products
* Males who are sexually active and not surgically sterilised (vasectomy or otherwise) and their partners that are not using a highly effective contraception method, from randomisation until 90 days after dosing, such as double barrier contraception (e.g. condom and spermicide) or combination of either an oral ontraceptive, a contraceptive patch, a diaphragm or intrauterine device, together with a physical barrier such as condom. Male subjects must also agree to refrain from sperm donation from randomisation until 90 days after last dosing
* Female who is pregnant, breast-feeding or intends to become pregnant or is of child-bearing potential and not using adequate contraceptive methods (adequate contraceptive measures as required by local regulation or practice) (adequate contraceptive measures are defined as sterilisation, hormonal intrauterine device, oral contraceptives, condom with spermicide sexual abstinence or vasectomised partner)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2016-10-19 (Actual); Primary Completion 2017-06-17 (Actual); Study Completion 2017-07-04 (Actual)

PRIMARY OUTCOMES:
The ratio of suppression of endogenous glucose production relative to total glucose lowering effect | Two weeks of treatment

SECONDARY OUTCOMES:
Number of treatment emergent adverse events | Time of first trial product administration to 7 days (7 times 24 hours) after last trial product administration

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Graz, Austria